CLINICAL TRIAL: NCT03353389
Title: Review of Trend in Incidence and Characteristics of Hospital-acquired Acute Kidney Injury in Hospital Selayang
Acronym: HA-AKI-HS
Status: Completed | Type: Observational
Sponsor: Selayang Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HA-AKI-1
Record Dates: First submitted 2017-11-18; First posted 2017-11-27 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury; Acute Renal Failure; Kidney Failure, Acute; Hospital Acquired Condition
Keywords: Acute Kidney Injury; Hospital-acquired Acute Kidney Injury; Community-acquired Acute Kidney Injury; Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury; Iatrogenic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No AKI: Adult admissions without Acute Kidney Injury during their stay
  Interventions: Other: No AKI
- CA-AKI: Adult admissions with Acute Kidney Injury diagnosed within 48 hours during their stay (Community-acquired Acute Kidney Injury)
  Interventions: Other: CA-AKI
- HA-AKI: Adult admissions with Acute Kidney Injury diagnosed after 48 hours during their stay (Hospital-acquired Acute Kidney Injury)
  Interventions: Other: HA-AKI

INTERVENTIONS:
Other: No AKI — Subjects will be allocated into this group if they did not acquire Acute Kidney Injury during admission.
  Groups: No AKI
Other: CA-AKI — CA-AKI is defined by any patient who developed AKI (as per definition below) within 48 hours of hospital admission.
  Definition of AKI:
  i. An increase in serum creatinine of 0.3 mg/dl (26.5 μmol/l) within 48 hours OR ii. An increase in serum creatinine to more or equal to 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days
  Definition for baseline creatinine:
  i. The baseline creatinine level is defined as the creatinine level at or within 7 days before the hospital admission, OR ii. at the hospital admission OR iii. the lowest creatinine (excluding the post dialysis creatinine if dialysis is initiated) during the index hospitalisation for those whose baseline creatinine were unknown.
  Groups: CA-AKI
Other: HA-AKI — HA-AKI is defined by any patient who developed AKI (as per definition below) after 48 hours of hospital admission.
  Definition of AKI:
  i. An increase in serum creatinine of 0.3 mg/dl (26.5 μmol/l) within 48 hours OR ii. An increase in serum creatinine to more or equal to 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days
  Definition for baseline creatinine:
  i. The baseline creatinine level is defined as the creatinine level at or within 7 days before the hospital admission, OR ii. at the hospital admission OR iii. the lowest creatinine (excluding the post dialysis creatinine if dialysis is initiated) during the index hospitalisation for those whose baseline creatinine were unknown.
  Groups: HA-AKI

SUMMARY:
This retrospective cohort study aims to investigate the incidence, risk factors and outcomes of Hospital-acquired Acute Kidney Injury in Hospital Selayang, a tertiary hospital at Malaysia, over 15 years.

DETAILED DESCRIPTION:
This is a retrospective cohort study involving 5-yearly trend from 2002 to 2017 for analysis. Laboratory serum creatinine (SCr) results of all patients admitted during study period will be retrieved from the hospital Laboratory Information System. A preliminary screening list will be generated by using STATA program from the SCr results. The nephrologist will then determine HA-AKI and CA-AKI as per inclusion and exclusion criteria. Data collectors will collect all relevant data from these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult admissions to Hospital Selayang from

  * 1st July 2001 to 30th June 2002
  * 1st July 2006 to 30th June 2007
  * 1st July 2011 to 30th June 2012
  * 1st July 2016 to 30th June 2017

Exclusion Criteria:

* End Stage Renal Failure and on Renal Replacement Therapy (Hemodialysis, peritoneal dialysis or Renal Transplant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult admissions to Hospital Selayang from
  * 1st July 2001 to 30th June 2002
  * 1st July 2006 to 30th June 2007
  * 1st July 2011 to 30th June 2012
  * 1st July 2016 to 30th June 2017
Sampling Method: Non-Probability Sample
Enrollment: 170000 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Hospital-acquired Acute Kidney Injury | During admissions to study site (Year 2001-2002, Year 2006-2007, Year 2011-2012, Year 2016-2017)
  Incidence of Hospital-acquired Acute Kidney Injury among the adult admissions

SECONDARY OUTCOMES:
Renal Recovery from Hospital-acquired Acute Kidney Injury | 90 days after diagnosis of Acute Kidney Injury
  Renal Recovery among adult admissions for Hospital-acquired Acute Kidney Injury
In-hospital Mortality from Hospital-acquired Acute Kidney Injury | During admissions to study site with Hospital-acquired Acute Kidney Injury, through study completion (an average of 1 year)
  Mortality rate among adult admissions for Hospital-acquired Acute Kidney Injury

CONTACTS AND LOCATIONS:
Overall Officials: Lee Fei Yee, BPharm, Principal Investigator — Clinical Research Centre
Locations (1):
- Selayang Hospital, Batu Caves, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
Subject's names will be kept on a password-protected database and will be linked only with a study identification number for this research. The identification number instead of patient identifiers will be used on subject data sheets. All data will be entered into a computer that is password protected. On completion of study, data in the computer will be copied to CDs and the data in the computer erased. CDs and any hardcopy data will be stored in a locked office of the investigators and maintained for a minimum of three years after the completion of the study. The CDs and data will be destroyed after that period of storage. No personal information will be disclosed and subjects will not be identified when the findings of the survey are published.

REFERENCES:
- [Result] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Result] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Result] Kumar S, Raina S, Vikrant S, Patial RK. Spectrum of acute kidney injury in the Himalayan region. Indian J Nephrol. 2012 Sep;22(5):363-6. doi: 10.4103/0971-4065.103914. PMID 23326047
- [Result] Jannot AS, Burgun A, Thervet E, Pallet N. The Diagnosis-Wide Landscape of Hospital-Acquired AKI. Clin J Am Soc Nephrol. 2017 Jun 7;12(6):874-884. doi: 10.2215/CJN.10981016. Epub 2017 May 11. PMID 28495862
- [Result] Cely JE, Mendoza EJ, Olivares CR, Sepulveda OJ, Acosta JS, Baron RA, Diaztagle JJ. Incidence and Risk Factors for Early Acute Kidney Injury in Nonsurgical Patients: A Cohort Study. Int J Nephrol. 2017;2017:5241482. doi: 10.1155/2017/5241482. Epub 2017 Apr 11. PMID 28487772
- [Result] Swaminathan M, Hudson CC, Phillips-Bute BG, Patel UD, Mathew JP, Newman MF, Milano CA, Shaw AD, Stafford-Smith M. Impact of early renal recovery on survival after cardiac surgery-associated acute kidney injury. Ann Thorac Surg. 2010 Apr;89(4):1098-104. doi: 10.1016/j.athoracsur.2009.12.018. PMID 20338313
- [Result] Rewa O, Bagshaw SM. Acute kidney injury-epidemiology, outcomes and economics. Nat Rev Nephrol. 2014 Apr;10(4):193-207. doi: 10.1038/nrneph.2013.282. Epub 2014 Jan 21. PMID 24445744
- [Result] Nash K, Hafeez A, Hou S. Hospital-acquired renal insufficiency. Am J Kidney Dis. 2002 May;39(5):930-6. doi: 10.1053/ajkd.2002.32766. PMID 11979336
- [Result] Hou SH, Bushinsky DA, Wish JB, Cohen JJ, Harrington JT. Hospital-acquired renal insufficiency: a prospective study. Am J Med. 1983 Feb;74(2):243-8. doi: 10.1016/0002-9343(83)90618-6. PMID 6824004
- [Result] Ali T, Khan I, Simpson W, Prescott G, Townend J, Smith W, Macleod A. Incidence and outcomes in acute kidney injury: a comprehensive population-based study. J Am Soc Nephrol. 2007 Apr;18(4):1292-8. doi: 10.1681/ASN.2006070756. Epub 2007 Feb 21. PMID 17314324

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT03353389/Prot_SAP_000.pdf